CLINICAL TRIAL: NCT03988686
Title: Zhongshan Hospital, Fudan University
Brief Title: Testing Radical Prostatectomy in Chinese Men With Prostate Cancer and oligoMetastases to the Bone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: University College, London (Other)
Responsible Party: Principal Investigator, Jianming Guo, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2019-065
Record Dates: First submitted 2019-06-08; First posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Prostate Cancer Metastatic
Keywords: oligometastasis; prostate cancer; radical prostatectomy; progression-free survival; quality of life
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Radical prostatectomy plus standard care
  Interventions: Procedure: Radical prostatectomy plus standard care; Drug: Standard of care for metastatic prostate cancer
- Comparator Group (Active Comparator): Standard care, currently ADT +/- other systemic therapies.
  Interventions: Drug: Standard of care for metastatic prostate cancer

INTERVENTIONS:
Procedure: Radical prostatectomy plus standard care — To add radical prostatectomy on the basis of current standard of care for those with oligometastatic prostate cancer
  Arms: Intervention Group
Drug: Standard of care for metastatic prostate cancer — androgen deprivation therapy with or without other systemic therapies based on current guidelines for metastatic prostate cancer

SUMMARY:
This study is to examine whether radical prostatectomy can impact survival and quality-of-life in men with oligo-metastatic prostate cancer.

DETAILED DESCRIPTION:
In this study, patients with oligo-metastatic prostate cancer will be randomized to radical prostatectomy plus standard care and standard care only. Standard care refers to androgen deprivation therapy (ADT) +/- other systemic therapies. Time to disease progression and post-treatment quality of life will be assessed and compared.

ELIGIBILITY:
Inclusion Criteria:

* Participants is willing and able to give informed consent for participation in the study
* Male aged 19-75 years.
* Diagnosed with oligo-metastatic prostate cancer (1-3 skeletal lesions on bone specific imaging, no visceral metastases).
* Locally resectable tumor (clinical/radiological stage T1-T3).
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Suitable for radical prostatectomy within 12 months of starting standard care.

Exclusion Criteria:

* Contraindications to radical prostatectomy.
* Visceral metastases.
* Prior radiotherapy to the abdomen/pelvis or to skeletal metastases.
* Any systemic therapy of prostate cancer (including standard care) for 12 or more months prior to enrollment.
* Current involvement in other interventional research.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
the time to castrate resistance | 36 months after randomization
  The time to treatment failure defined as castrate resistance will be recorded via routine patient follow-up interviews.

SECONDARY OUTCOMES:
Quality of life in patients post-randomization | three month post randomization
  EuroQOL 5 dimensions 5 levels (EQ-5D-5L) questionnaire will be used to assess quality of life in patients after randomization with different treatments. This is designed to measure health-related quality of life. It consists of a questionnaire and a visual analogue scale. The subjects in 5 dimensions i.e. mobility, self-care, usual activities, pain/discomfort and anxiety/depression are asked to grade their own current level of function in each dimension into one of five levels of disability (i.e. I have no problems waling about, slight problems, moderate problems, severe problems, or unable to walk). This tool also has an overall health scale where the rater selects a number between 1-100 to describe the condition of their health, 100 being the best imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Ming Guo, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China